CLINICAL TRIAL: NCT07018115
Title: The Effect of Preoperative Patient Information Strategies on Anxiety and Hemodynamic Responses During Third Molar Extraction
Brief Title: Anxiety and Hemodynamic Changes in Third Molar Extraction After Patient Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ummugulsum Coskun (Other)
Responsible Party: Sponsor-Investigator, Ummugulsum Coskun, Assistant Professor of Oral and Maxillofacial Surgery, DDS, PhD, Altinbas University
Organization: Altinbas University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015/30
Record Dates: First submitted 2025-05-25; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Dental Anxiety; Hemodynamic; Molar, Third; Tooth Extraction; Tooth Impacted
Keywords: Dental Anxiety; Patient Education; Impacted Third Molar; Pain Management; Hemodynamic Changes
MeSH Terms: conditions — Tooth, Impacted; Agnosia | interventions — Carticaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: This randomized, parallel assignment clinical trial allocates participants into three independent groups to compare the effects of different preoperative patient information strategies (basic explanation, detailed verbal explanation, visual animation) on anxiety levels and physiological responses during third molar extraction. Each group receives only its assigned type of information, and outcomes are measured and compared separately across the groups.
Masking Description: Due to the nature of the interventions, which involved providing different types of preoperative patient education (basic explanation, detailed verbal explanation, visual animation), masking was not feasible, and both participants and investigators were aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Other): Participants receive only a basic, brief explanation of the surgical procedure without additional detailed verbal or visual information.
  Interventions: Other: Basic Preoperative Information; Drug: Articaine 4% with epinephrine 1:100,000; Procedure: Surgical extraction of impacted mandibular third molar; Device: Multiparameter patient monitor
- Verbal Information Group (Experimental): Participants receive a comprehensive verbal explanation of the surgical procedure, covering all key steps such as anesthesia, incision, bone removal, tooth sectioning, and suturing, delivered in clear, non-technical language to optimize patient understanding.
  Interventions: Other: Detailed Verbal Preoperative Information; Drug: Articaine 4% with epinephrine 1:100,000; Procedure: Surgical extraction of impacted mandibular third molar; Device: Multiparameter patient monitor
- Visual Information Group (Experimental): Participants receive the same detailed verbal explanation as the verbal information group, supplemented with a 2D animated video illustrating the surgical procedure
  Interventions: Other: Visual Preoperative Information (2D Animation); Drug: Articaine 4% with epinephrine 1:100,000; Procedure: Surgical extraction of impacted mandibular third molar; Device: Multiparameter patient monitor

INTERVENTIONS:
Other: Basic Preoperative Information — Participants receive a brief, non-detailed explanation of the surgical procedure.
  Other Names: Control Information; Minimal Explanation
  Arms: Control Group
Other: Detailed Verbal Preoperative Information — Participants receive a detailed verbal explanation covering the surgical procedure, including anesthesia, incision, bone removal, tooth sectioning, and suturing.
  Other Names: Verbal Explanation; Detailed Verbal Education; Verbal Counseling
  Arms: Verbal Information Group
Other: Visual Preoperative Information (2D Animation) — Participants receive a 2D animated video illustrating the surgical procedure in addition to the detailed verbal explanation.
  Other Names: Animated Video; Visual Education; Animation-Based Information
  Arms: Visual Information Group
Drug: Articaine 4% with epinephrine 1:100,000 — A local anesthetic solution (Ultracain D-S; Aventis) administered in a dose of 2 ml for all patients. The anesthetic was injected to achieve regional nerve block anesthesia (inferior alveolar, lingual, and buccal nerves) prior to the surgical extraction of impacted mandibular third molars. The solution contains epinephrine as a vasoconstrictor to prolong anesthetic effect and minimize intraoperative bleeding.
Procedure: Surgical extraction of impacted mandibular third molar — A standardized surgical protocol was followed for the removal of impacted mandibular third molars. All procedures were performed under local anesthesia using a mucoperiosteal flap approach. The surgery included a linear or triangular incision, elevation of the mucoperiosteal flap, ostectomy using rotary instruments as needed, and tooth sectioning in cases of difficult extraction. The socket was irrigated with sterile saline solution, and hemostasis was achieved. Wound closure was performed with 4.0 silk sutures. All surgeries were conducted by experienced oral and maxillofacial surgeons without sedation or premedication. The entire procedure was monitored for hemodynamic parameters including heart rate, blood pressure, and oxygen saturation.
Device: Multiparameter patient monitor — A hospital-grade multiparameter monitor was used to measure and record patients' vital signs at five defined surgical stages: before surgery, after information delivery, after local anesthesia, during tooth extraction, and postoperatively. The monitor continuously recorded heart rate (HR), systolic and diastolic blood pressure (SBP and DBP), and peripheral oxygen saturation (SpO₂). The collected data were used to evaluate physiological responses associated with anxiety and surgical stress.

SUMMARY:
This randomized clinical trial investigates the effect of different preoperative patient information strategies on anxiety levels and hemodynamic responses during third molar extraction. Ninety-seven patients were assigned to control, verbal information, or visual (animation) information groups. Anxiety was measured using the Modified Dental Anxiety Scale (MDAS) and State-Trait Anxiety Inventory (STAI), while heart rate, blood pressure, oxygen saturation, and pain were recorded. The study aims to assess whether educational interventions can reduce anxiety and improve patient comfort during oral surgery.

DETAILED DESCRIPTION:
This prospective, randomized clinical trial was designed to evaluate the effect of different preoperative patient information strategies on anxiety levels, hemodynamic responses, and pain perception during the surgical extraction of impacted mandibular third molars. Third molar extraction is a common procedure in oral and maxillofacial surgery, often associated with elevated patient anxiety, which can negatively affect both psychological well-being and physiological parameters such as heart rate and blood pressure.

In this study, 97 patients requiring surgical removal of a single impacted mandibular third molar were recruited and randomly assigned into one of three groups:

1. Control group - provided with a brief, basic explanation of the surgical procedure;
2. Verbal information group - provided with a detailed, non-technical verbal explanation covering the anesthesia, surgical steps, and post-operative care;
3. Visual information group - provided with the same verbal explanation plus an educational 2D animation illustrating the surgical process.

The anxiety levels of participants were measured using two validated scales: the Modified Dental Anxiety Scale (MDAS) and the State-Trait Anxiety Inventory (STAI), both before and after surgery. Physiological measurements, including heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), and oxygen saturation (SaO₂), were recorded at five standardized time points: before surgery, after information delivery and before anesthesia, after anesthesia, during tooth extraction, and in the postoperative period. Pain levels were assessed during the procedure using a Visual Analog Scale (VAS).

All surgeries were conducted under local anesthesia by experienced oral surgeons, following a standardized surgical protocol to minimize operator-related variability. The study also considered demographic and clinical variables, such as patient age, sex, education level, and the depth of impaction of the third molar, as potential factors influencing anxiety and physiological responses.

The study was conducted at the Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Karadeniz Technical University, and received approval from the university's ethics committee (approval number 2015/30). The primary hypothesis was that providing patients with detailed verbal or visual information would reduce preoperative anxiety compared to basic explanations, and that visual tools might offer additional benefits by enhancing patient understanding and comfort.

The results demonstrated that while anxiety scores generally decreased postoperatively across all groups, the visual (animation) information group showed significantly better oxygen saturation levels during extraction and in the postoperative period, suggesting a positive physiological impact. However, no significant differences were found between groups regarding pain scores or overall surgical duration.

These findings highlight the importance of preoperative patient education and suggest that incorporating visual educational tools, such as animations, may improve physiological stability and patient experience during oral surgical procedures. Further research is warranted to refine these strategies and explore their long-term benefits in various dental and surgical contexts.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Requiring surgical removal of a impacted mandibular third molar
* Ability to read and complete the questionnaires
* Willingness to participate in the study

Exclusion Criteria:

* Age < 18 years
* History of systemic disease contraindicating surgery
* Poor oral hygiene
* Current pericoronitis or acute infection around the third molar
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-02-10 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Modified Dental Anxiety Scale (MDAS) Score After Third Molar Surgery | From baseline (before patient education) to within 1 hour after completion of third molar extraction
  The Modified Dental Anxiety Scale (MDAS) is a validated questionnaire consisting of 5 items, each scored from 1 (not anxious) to 5 (extremely anxious), producing a total score range of 5 to 25. Higher scores indicate higher levels of dental anxiety. In this study, participants completed the MDAS before receiving any information (preoperative baseline) and again immediately after third molar extraction (postoperative). The change in MDAS score from baseline to postoperative was calculated to assess the effect of patient education interventions on dental anxiety levels.
Change from Baseline in Spielberger State-Trait Anxiety Inventory (STAI-Trait) Score After Third Molar Surgery | From baseline (before patient education) to within 1 hour after completion of third molar extraction
  The Spielberger State-Trait Anxiety Inventory - Trait (STAI-T) subscale is a validated self-reported questionnaire with 20 items, each rated from 1 (almost never) to 4 (almost always), giving a total score between 20 and 80. Higher scores indicate higher levels of trait anxiety. In this study, participants completed the STAI-T before receiving any information (preoperative baseline) and again immediately after third molar extraction (postoperative). The change in STAI-Trait score from baseline to postoperative was calculated to assess the effect of patient education on trait anxiety.
Change from Baseline in Spielberger State-Trait Anxiety Inventory (STAI-State) Score After Third Molar Surgery | From baseline (before patient education) to within 1 hour after completion of third molar extraction
  The Spielberger State-Trait Anxiety Inventory - State (STAI-S) subscale is a validated self-reported questionnaire with 20 items, each rated from 1 (not at all) to 4 (very much so), giving a total score between 20 and 80. Higher scores indicate higher levels of state anxiety. In this study, participants completed the STAI-S before receiving any information (preoperative baseline) and again immediately after third molar extraction (postoperative). The change in STAI-State score from baseline to postoperative was calculated to assess the effect of patient education on state anxiety.

SECONDARY OUTCOMES:
Change in Heart Rate (HR) During Third Molar Surgery | From 10 minutes before local anesthesia to 10 minutes after completion of surgery (total duration approximately 30 minutes)
  Heart rate was measured in beats per minute (bpm) at five predefined time points:
  T1: 10 minutes before surgery (baseline), T2: 5 minutes after patient education and immediately before local anesthesia, T3: 5 minutes after local anesthesia administration, T4: At the moment of tooth removal (typically between minutes 12 and 20 of the procedure), T5: 10 minutes after completion of surgery and suturing. Changes in heart rate across these phases were analyzed to evaluate the physiological impact of surgical stress and preoperative patient information.
Change in Systolic Blood Pressure (SBP) During Third Molar Surgery | From 10 minutes before local anesthesia to 10 minutes after completion of surgery (total duration approximately 30 minutes)
  Systolic blood pressure (SBP) was measured at five predefined time points:
  T1: 10 minutes before surgery (baseline), T2: 5 minutes after patient education and immediately before local anesthesia, T3: 5 minutes after local anesthesia administration, T4: At the moment of tooth removal (typically between minutes 12 and 20 of the procedure), T5: 10 minutes after completion of surgery and suturing. Changes in SBP were analyzed to assess physiological responses to preoperative patient education and surgical stress.
Change in Diastolic Blood Pressure (DBP) During Third Molar Surgery | From 10 minutes before local anesthesia to 10 minutes after completion of surgery (total duration approximately 30 minutes)
  Diastolic blood pressure (DBP) was measured in mmHg at five predefined time points:
  T1: 10 minutes before surgery (baseline), T2: 5 minutes after patient education and immediately before local anesthesia, T3: 5 minutes after local anesthesia administration, T4: At the moment of tooth removal (typically between minutes 12 and 20 of the procedure), T5: 10 minutes after completion of surgery and suturing. These measurements were used to assess physiological stress responses during third molar surgery and the potential influence of preoperative patient education.
Change in Peripheral Oxygen Saturation (SpO₂) During Third Molar Surgery | From 10 minutes before local anesthesia to 10 minutes after completion of surgery (total duration approximately 30 minutes)
  Peripheral oxygen saturation (SpO₂) was measured as a percentage (%) at five predefined time points:
  T1: 10 minutes before surgery (baseline), T2: 5 minutes after patient education and immediately before local anesthesia, T3: 5 minutes after local anesthesia administration, T4: At the moment of tooth removal (typically between minutes 12 and 20 of the procedure), T5: 10 minutes after completion of surgery and suturing. These measurements were analyzed to identify potential changes in oxygen saturation associated with surgical stress and the impact of different patient education methods.
Pain Intensity During Tooth Extraction Measured by Visual Analog Scale (VAS) | From the start of tooth elevation to immediately after tooth removal (approximately minutes 15 to 20 of the procedure)
  Pain was assessed using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst possible pain). Patients were asked to report their pain level immediately after the tooth was extracted, while still in the surgical setting. This measure reflects the intensity of pain experienced specifically at the moment of tooth removal and was used to evaluate its relationship with the type of preoperative patient education provided.
Duration of Third Molar Extraction Procedure | From the first surgical incision to the final suture placement (approximately 10 to 30 minutes total)
  The duration of the surgical procedure was recorded in minutes, starting with the first incision and ending with the placement of the final suture. This variable was used to evaluate whether the type of preoperative patient education influenced the total procedure time or surgical efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Ummugulsum Coskun, DDS, PhD, Principal Investigator — Altinbas University

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available to qualified researchers upon reasonable request after publication of the study results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The individual participant data (IPD) and supporting information will be available upon publication of the study results and will remain available for 5 years thereafter.
Access Criteria: Qualified researchers can request IPD, protocol, and analysis plan by contacting the corresponding author. Data will be shared under a data use agreement after review.